CLINICAL TRIAL: NCT04378205
Title: Pulpal Blood Flow Changes Related to Using SuperElastic 0.018-inch Nickel Titanium as the First Orthodontic Alignment Archwire: A Prospective Clinical Trial
Brief Title: Pulpal Blood Flow Changes Using SuperElastic 0.018-inch Nickel Titanium
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Jordan University of Science and Technology (Other)
Responsible Party: Principal Investigator, Elham Abu Alhaija, Professor, Jordan University of Science and Technology
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 39/2018
Record Dates: First submitted 2020-05-02; First posted 2020-05-07 (Actual); Last update posted 2020-05-07 (Actual); Status verified 2020-05

CONDITIONS: Orthodontic Appliance
Keywords: Pulpal blood flow; Pfixed appliance; Alignment arch wire

STUDY DESIGN:
Intervention Model Description: A split mouth study design was applied. Each patient received 2 archwire sizes at one time joined in the midline by crimpable hook and applied in the lower arch. Patients were assigned into one of 2 groups based on archwire sizes used. Group 1:- 0.014-inch and 0.018-inch NiTi Group 2:- 0.016-inch and 0.018-inch NiTi.
Who Masked: Participant, Outcomes Assessor
Masking Description: Psarticipants did not know which size is allocated/side.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 0.014/0.018 NiTi arch wire (Experimental): 0.014-inch NiTi on one side /0.018-inch NiTi on the other side (Nitinol SuperElastic 3M, Unitek) for initial alignment. This group included 20 patients
  Interventions: Procedure: 0.014-inch NiTi on one side /0.018-inch NiTi on the other side
- 0.016/0.018 NiTi arch wire (Experimental): 0.016-inch NiTi on one side / 0.018-inch NiTi on the other side (Nitinol SuperElastic 3M, Unitek) for initial alignment. This group included 20 patients
  Interventions: Procedure: 0.016-inch NiTi on one side /0.018-inch NiTi on the other side

INTERVENTIONS:
Procedure: 0.014-inch NiTi on one side /0.018-inch NiTi on the other side — Where each patient received 2 archwire sizes (0.014-inch and 0.018-inch) at one time joined in the midline by crimpable hook and applied in the lower arch.
  Arms: 0.014/0.018 NiTi arch wire
Procedure: 0.016-inch NiTi on one side /0.018-inch NiTi on the other side — Where each patient received 2 archwire sizes (0.016-inch and 0.018-inch) at one time joined in the midline by crimpable hook and applied in the lower arch.
  Arms: 0.016/0.018 NiTi arch wire

SUMMARY:
to record pulpal blood flow (PBF) changes associated with using 0.018-inch Nickel Titanium (NiTi) as the first alignment archwire during fixed orthodontic treatment.

DETAILED DESCRIPTION:
Forty healthy patients with lower arch mild crowding with less than 2mm contact point displacement at any teeth were included. A split mouth study design was applied. Where each patient received 2 archwire sizes at one time joined in the midline by crimpable hook and applied in the lower arch.

Patients were assigned into one of 2 groups based on archwire sizes used. Group (1); 0.014-inch and 0.018-inch NiTi and Group (2); 0.016-inch and 0.018-inch NiTi. A Laser Doppler Flowmeter was used to measure PBF at different time intervals (T0-T5).

ELIGIBILITY:
Inclusion Criteria:

* age 18-25 years
* Class I skeletal malocclusion
* Mild lower arches crowding.
* Contact point displacement less than 2 mm.
* No previous orthodontic treatment

Exclusion Criteria:

* Missing teeth
* Poor oral hygiene
* deep carious teeth
* history of previous trauma
* any medical conditions affecting blood vessels
* smokers

Ages: 18 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2018-09-01 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
Pulpal blood flow changes | up to 4 weeks
  Measurements were taken by the use of Laser Doppler Flowmeter mm/s

CONTACTS AND LOCATIONS:
Overall Officials: Elham Abu Alhaija, PhD, Principal Investigator — Jordan University of Science and Technology
Locations (1):
- Dental Faculty/Jordan university of Science and Technology Dental Teaching Clinics, Irbid, Jordan

IPD SHARING:
Plan to Share IPD: No